CLINICAL TRIAL: NCT07264725
Title: Multiple Sclerosis Care in a Conflict-Affected Health System: Diagnostic Delay, Treatment Access, and Disability Outcomes in Libya
Brief Title: Libyan Multiple Sclerosis Registry Study
Status: Completed | Type: Observational
Sponsor: University of Zintan (Other)
Responsible Party: Sponsor
Other Study IDs: ZFM-2024-MS03; ZFM/2024/MS-03 (Registry Identifier: Libyan Multiple Sclerosis Registry)
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis MS Relapsing-Remitting MS Secondary Progressive MS Primary Progressive MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Disease-Modifying Therapies — This is an observational study. No medications are assigned, administered, or modified by the study team. Disease-modifying therapies (DMTs) are recorded only as exposure variables based on routine clinical care. All drugs listed in this record are prescribed independently by treating neurologists as part of standard care, and the study does not influence treatment decisions in any way.

SUMMARY:
This study aims to understand differences in access to diagnosis and treatment for people with multiple sclerosis (MS) receiving care in Libya. The study uses data from the Libyan Multiple Sclerosis Registry, which collects clinical and treatment information from patients at two tertiary neurology centres. The main focus is to examine how long it takes for patients to receive an MS diagnosis, who has access to high-efficacy disease-modifying therapies, and how these factors relate to disability levels. The results will help identify gaps in MS care within a conflict-affected health system and guide improvements in services for patients in Libya.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosis of multiple sclerosis according to the 2017 McDonald criteria
* Receiving care at Tripoli University Hospital or Omar Askar Hospital
* Able to provide written informed consent
* Recorded EDSS score at registry entry
* Availability of core demographic and diagnostic information

Exclusion Criteria:

* Clinically isolated syndrome (CIS)
* Age younger than 18 years
* Absence of confirmed multiple sclerosis diagnosis
* Missing key clinical variables required for primary analysis (EDSS, phenotype, or DMT information)
* Declined or unable to provide informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with multiple sclerosis receiving neurological care at two tertiary centres in western Libya: Tripoli University Hospital in Tripoli and Omar Askar Hospital in Zliten. Patients are enrolled into the Libyan Multiple Sclerosis Registry during routine clinical visits, with disability assessments and treatment information recorded by trained neurologists. The study population reflects a broad range of MS phenotypes, socioeconomic backgrounds, and treatment exposures within a conflict-affected health system.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Moderate-to-Severe Disability (EDSS ≥3.0) | At registry entry
  Disability measured using the Expanded Disability Status Scale (EDSS). Moderate-to-severe disability is defined as EDSS ≥3.0, assessed by trained neurologists using standardised procedures.
Moderate-to-Severe Disability (EDSS ≥3.0) | At registry entry

SECONDARY OUTCOMES:
EDSS Ordinal Disability Categories | At registry entry
  Disability severity categorised using the Expanded Disability Status Scale (EDSS) into three groups:
  0-2.5 (mild), 3.0-5.5 (moderate), and ≥6.0 (severe). EDSS scores are assessed by trained neurologists at the time of registry entry.

CONTACTS AND LOCATIONS:
Locations (1):
- Tripoli University Hospital, Zintan, Libya

IPD SHARING:
Plan to Share IPD: No